CLINICAL TRIAL: NCT04415658
Title: A Multicenter Randomized Placebo-Controlled Trial of Intravenous Thyroxine for Heart-Eligible Brain Dead Organ Donors
Brief Title: Intravenous Thyroxine for Heart-Eligible Organ Donors
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Mid-America Transplant (Other)
Responsible Party: Principal Investigator, Rajat Dhar, Professor, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ODRC-002
Record Dates: First submitted 2020-05-27; First posted 2020-06-04 (Actual); Results first posted 2024-01-10 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2023-12

CONDITIONS: Brain Death; Heart Failure
Keywords: Organ donor
MeSH Terms: conditions — Brain Death; Heart Failure | interventions — Thyroxine; Sodium Chloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Thyroxine (Experimental): Intravenous thyroxine infusion
  Interventions: Drug: Thyroxine
- Saline Placebo (Placebo Comparator): Intravenous saline infusion
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Thyroxine — Infusion prepared by mixing 500 μg of drug in 500-ml of normal saline (i.e. concentration of 1 μg/ml) and enclosing the bag in an opaque sleeve. Infusion started at 30 μg/hour (30 ml/hour) for twelve hours.
  Arms: Thyroxine
Drug: Saline — The placebo will be a 500-ml bag of normal saline (without active drug) also enclosed in an opaque sleeve. This infusion will also be started at 30 ml/hour for twelve hours.
  Arms: Saline Placebo

SUMMARY:
This randomized controlled trial will evaluate whether intravenous thyroxine infusion given to brain-dead organ donors who are eligible to donate hearts for 12 hours will result in more hearts transplanted than saline placebo

DETAILED DESCRIPTION:
Background: Brain death frequently induces hemodynamic instability and cardiac stunning. Impairments in cardiac performance are major contributors to hearts from otherwise eligible organ donors not being transplanted. Deficiencies in pituitary hormones (including thyroid stimulating hormone) may contribute to hemodynamic instability and replacement of thyroid hormone has been proposed as a means of improving stability and increasing hearts available for transplantation. Intravenous thyroxine is commonly used in donor management. However, small controlled trials have not been able to demonstrate efficacy.

Methods: This multicenter study will involve organ procurement organizations (OPOs) across the country. A total of 800 heart-eligible brain dead organ donors who require vasopressor support will be randomly assigned to intravenous thyroxine for at least 12-hours or saline placebo. The primary study hypothesis is that thyroxine treatment results in more hearts transplanted. Additional outcome measures are time to achieve hemodynamic stability (weaning off vasopressors) and improvement in cardiac ejection fraction on echocardiography.

Discussion: This will be the largest randomized controlled study to evaluate the efficacy of thyroid hormone treatment for organ donor management. By collaborating across multiple OPOs, it will be able to enroll an adequate number of donors and be powered to definitively answer the critical question of whether treatment increases hearts transplanted and/or provides other hemodynamic benefits.

ELIGIBILITY:
Inclusion Criteria:

* Declared dead by neurologic criteria (brain dead)
* Authorization for organ donation and research
* On one or more vasopressors and/or inotropes

Exclusion Criteria:

* Brain death declared more than 24 hours prior
* Only vasopressor is vasopressin
* Weight < 45 kg (100 lbs)
* Known coronary artery disease or history of myocardial infarction
* Known valvular heart disease
* Prior sternotomy or cardiac surgery
* Donor at VA hospital
* Received intravenous or oral thyroxine within past month
* Known HIV+ status
* Other reason donor is unable to receive study drug (determined by on-site personnel)

Ages: 14 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 838 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2022-11-06 (Actual); Study Completion 2022-12-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rajat Dhar, MD, Principal Investigator — Washington University School of Medicine
Locations (14):
- United States (14):
  - Donor Network of Arizona, Phoenix, Arizona
  - Lifesharing, San Diego, California
  - Donor Alliance, Denver, Colorado
  - OurLegacy, Maitland, Florida
  - Iowa Donor Network, North Liberty, Iowa
  - Midwest Transplant Network, Westwood, Kansas
  - Louisiana Organ Procurement Agency, Covington, Louisiana
  - Mid-America Transplant Services, St Louis, Missouri
  - Lifebanc, Cleveland, Ohio
  - LifeShare of Oklahoma, Oklahoma City, Oklahoma
  - Southwest Transplant Alliance, Dallas, Texas
  - Texas Organ Sharing Alliance, San Antonio, Texas
  - DonorConnect, Murray, Utah
  - LifeCenter Northwest, Bellevue, Washington

IPD SHARING:
Plan to Share IPD: No
Researchers within the study consortium only

REFERENCES:
- [Background] Dhar R, Stahlschmidt E, Yan Y, Marklin G. A randomized trial comparing triiodothyronine (T3) with thyroxine (T4) for hemodynamically unstable brain-dead organ donors. Clin Transplant. 2019 Mar;33(3):e13486. doi: 10.1111/ctr.13486. Epub 2019 Feb 12. PMID 30689222
- [Background] Dhar R, Stahlschmidt E, Marklin G. A Randomized Trial of Intravenous Thyroxine for Brain-Dead Organ Donors With Impaired Cardiac Function. Prog Transplant. 2020 Mar;30(1):48-55. doi: 10.1177/1526924819893295. Epub 2019 Dec 5. PMID 31802716
- [Background] Dhar R, Marklin GF, Klinkenberg WD, Wang J, Goss CW, Lele AV, Kensinger CD, Lange PA, Lebovitz DJ. Intravenous Levothyroxine for Unstable Brain-Dead Heart Donors. N Engl J Med. 2023 Nov 30;389(22):2029-2038. doi: 10.1056/NEJMoa2305969. PMID 38048188
- [Derived] Dhar R, Klinkenberg D, Marklin G. A multicenter randomized placebo-controlled trial of intravenous thyroxine for heart-eligible brain-dead organ donors. Trials. 2021 Nov 27;22(1):852. doi: 10.1186/s13063-021-05797-2. PMID 34838132

RESULTS

PARTICIPANT FLOW:
Period: Initial Study Period (12 Hours)
Arm/Group | Thyroxine | Saline Placebo
Started | 419 | 419
Started Assigned Infusion | 411 | 384
Per-Protocol (Received assigned intervention for at least six hours) | 351 | 374
Cross-over (Crossed-over to other intervention within 12 hours) | 0 | 3
Stopped Infusion Early | 86 | 0
Completed (Refers to completing donor care, with organ allocation outcomes available) | 333 | 416
Not Completed | 86 | 3
Period: Open-Label (T4 Beyond 12 Hours)
Arm/Group | Thyroxine | Saline Placebo
Started (Total number of donors eligible to receive open-label) | 333 | 416
Completed (number who received thyroxine infusion beyond initial 12-hour study period) | 209 | 50
Not Completed | 124 | 366

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Thyroxine | Saline Placebo | Total
Number analyzed (Participants) | 419 | 419 | 838
Age, Continuous [Mean (Standard Deviation); unit: years] | 36 (11) | 36 (10) | 36 (10)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: missing data for 16 in T4 and 19 in NS group
  Participants
    number analyzed (Participants) | 403 | 400 | 803
    Female | 127 | 153 | 280
    Male | 276 | 247 | 523
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Missing data on 16 in T4 and 22 in NS group
  Participants
    White, non-Hispanic: number analyzed (Participants) | 403 | 397 | 800
    White, non-Hispanic | 252 | 278 | 530
    Black: number analyzed (Participants) | 403 | 397 | 800
    Black | 75 | 49 | 124
    Hispanic: number analyzed (Participants) | 403 | 397 | 800
    Hispanic | 60 | 63 | 123
    Asian, Pacific-Islander, other: number analyzed (Participants) | 403 | 397 | 800
    Asian, Pacific-Islander, other | 16 | 7 | 23
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 419 | 419 | 838
Blood Group [Count of Participants; unit: Participants]
  O | 224 | 214 | 438
  A | 134 | 148 | 282
  B | 50 | 49 | 99
  AB | 11 | 8 | 19
Cause of Death [Count of Participants; unit: Participants] — Population: missing demographic data for 16 in T4 and 22 in NS group
  Participants
    Anoxia: number analyzed (Participants) | 403 | 397 | 800
    Anoxia | 162 | 195 | 357
    Stroke / Cerebrovascular: number analyzed (Participants) | 403 | 397 | 800
    Stroke / Cerebrovascular | 87 | 79 | 166
    Trauma: number analyzed (Participants) | 403 | 397 | 800
    Trauma | 143 | 117 | 260
    Other: number analyzed (Participants) | 403 | 397 | 800
    Other | 11 | 6 | 17

OUTCOME MEASURES:

1. Primary Outcome: Heart Transplanted
Description: Whether heart is transplanted into living recipient
Time Frame: One week
Measure: Count of Participants; unit: Participants
Arm/Group | Thyroxine | Saline Placebo
Number analyzed (Participants) | 419 | 419
Participants | 230 | 223
Statistical Analysis 1: Comparison: Thyroxine vs Saline Placebo; 80% power to detect a 10% increase in hearts transplanted; Test type: Superiority; p = 0.57, Chi-squared, Corrected; Risk Ratio (RR) = 1.01, 95% CI 2-sided [0.97 to 1.07]

2. Primary Outcome: Graft Function
Description: 30-day graft survival of hearts transplanted from study donors, obtained from SRTR recipient registry
Time Frame: 30 days
Population: Only out of those hearts that were transplanted (not all study participants)
Measure: Count of Units; unit: hearts
Units Other Than Participants: hearts
Arm/Group | Thyroxine | Saline Placebo
Number analyzed (Participants) | 230 | 223
Number analyzed (hearts) | 230 | 223
hearts | 224 | 213
Statistical Analysis 1: Comparison: Thyroxine vs Saline Placebo; Non-inferiority analysis for thyroxine vs saline; Test type: Non-Inferiority — Six percent margin, assuming 96% graft survival in control group; p < 0.001, Regression, Logistic; Mean Difference (Final Values) = 1.9, 95% CI 2-sided [-2.3 to 6.0]

3. Secondary Outcome: Time Till Off Vasopressors
Description: Time in hours from randomization to when weaned off vasopressors (except vasopressin)
Time Frame: 72 hours
Population: out of those who began study infusion on vasopressors
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Thyroxine | Saline Placebo
Number analyzed (Participants) | 404 | 385
hours | 22 [19 to 31] | 25 [19 to 38]

4. Secondary Outcome: Weaned Off Vasopressors
Description: Weaned off vasopressors within twelve hours
Time Frame: 12 hours
Population: out of those who began the study infusion still on vasopressors (i.e. some had been weaned off prior to infusion)
Measure: Count of Participants; unit: Participants
Arm/Group | Thyroxine | Saline Placebo
Number analyzed (Participants) | 404 | 388
Participants | 143 | 152

5. Secondary Outcome: Time to Order Echo
Description: Time till hemodynamic stability permits ordering initial echocardiogram
Time Frame: 72 hours
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Thyroxine | Saline Placebo
Number analyzed (Participants) | 409 | 385
hours | 12 [11 to 13] | 13 [12 to 14]

6. Secondary Outcome: Ejection Fraction
Description: Left ventricular ejection fraction measured on first echocardiography
Time Frame: 72 hours
Population: only those who had echocardiography performed after study start
Measure: Mean (Standard Deviation); unit: percentage of ejection fraction
Arm/Group | Thyroxine | Saline Placebo
Number analyzed (Participants) | 350 | 336
percentage of ejection fraction | 59 (11) | 58 (12)

7. Secondary Outcome: Lungs Transplanted
Description: Whether the lungs were transplanted into a living recipient
Time Frame: 72 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Thyroxine | Saline Placebo
Number analyzed (Participants) | 419 | 419
Participants | 163 | 149

8. Other Pre Specified Outcome: Total Organs Transplanted
Description: Total number of organs transplanted (incl. lungs, liver, kidneys, heart, pancreas)
Time Frame: One week
Measure: Median (Inter-Quartile Range); unit: organs
Arm/Group | Thyroxine | Saline Placebo
Number analyzed (Participants) | 419 | 419
organs | 4 [3 to 5] | 4 [3 to 5]

ADVERSE EVENTS:
Time Frame: 1 week
Description: Serious adverse event defined as donor instability resulting in cardiac arrest or premature donor loss.
  Adverse events were collected for each arm combining all study periods, i.e. from study onset through end of donor management (organ recovery). These were not collected for each period (i.e. first 12 hours versus open-label period) separately.
Groups:
- Thyroxine: Intravenous thyroxine infusion
  Thyroxine: Infusion prepared by mixing 500 μg of drug in 500-ml of normal saline (i.e. concentration of 1 μg/ml) and enclosing the bag in an opaque sleeve. Infusion started at 30 μg/hour (30 ml/hour) for twelve hours.
  Donors were followed till organ recovery or end of management.
- Saline Placebo: Intravenous saline infusion
  Saline: The placebo will be a 500-ml bag of normal saline (without active drug) also enclosed in an opaque sleeve. This infusion will also be started at 30 ml/hour for twelve hours.
  Donors were followed till organ recovery or end of management.
Arm/Group | Thyroxine | Saline Placebo
All-Cause Mortality (participants affected / at risk) | 419/419 | 419/419
Serious Adverse Events (participants affected / at risk) | 2/419 | 3/419
Other Adverse Events (participants affected / at risk) | 51/419 | 16/419
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Thyroxine (N=419) | Saline Placebo (N=419)
Cardiac arrest / donor loss (Cardiac disorders) | 2 (2) | 3 (3) — Hemodynamic instability resulting in cardiac arrest and/or donor loss
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Thyroxine (N=419) | Saline Placebo (N=419)
Tachycardia (Cardiac disorders) | 16 (16) | 3 (3)
Hypertension (Cardiac disorders) | 26 (26) | 5 (5)
Atrial fibrillation (Cardiac disorders) | 7 (7) | 7 (7)
Ventricular ectopy (Cardiac disorders) | 5 (5) | 5 (5)
Ventricular tachycardia (Cardiac disorders) | 4 (4) | 1 (1) — not including unstable/leading to arrest
Misc/Other (General disorders) | 4 (4) | 2 (2) — includes rash, electrolyte disturbance, respiratory distress, pulmonary edema, hypotension

LIMITATIONS AND CAVEATS:
Not blinded, open-label use of levothyroxine permitted in control group after 12 hours (only 50 donors in that group received open-label, plus three who crossed-over to levothyroxine immediately after randomization)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol: Appendix (Data Forms) (2020-12-01): https://cdn.clinicaltrials.gov/large-docs/58/NCT04415658/Prot_003.pdf
  • Study Protocol and Statistical Analysis Plan: Study Protocol and SAP (2021-11-01): https://cdn.clinicaltrials.gov/large-docs/58/NCT04415658/Prot_SAP_005.pdf